CLINICAL TRIAL: NCT00688129
Title: KITS: School Readiness in Foster Care Efficacy Trial
Acronym: KITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Katherine C. Pears, Research Scientist, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: R01DA021424 (NIH); R01DA021424 (NIH)
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: School Readiness
Keywords: school readiness; foster care; maltreatment; literacy; social emotional skills; self regulation; caregiver involvement
MeSH Terms: conditions — Literacy; Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KITS Program (Experimental): The KITS intervention consists of: (a) child therapeutic play groups to facilitate the development of self-regulatory, social, and emergent literacy skills (2 times per week in summer, 1 times per week in the fall); (b) a bi-monthly psychoeducational support group to promote caregiver involvement in the child's emergent literacy and schooling and the use of effective parenting techniques; (c) home- and school-based behavioral consultation on an as needed basis.
  Interventions: Behavioral: KITS Program
- Services as usual (No Intervention)

INTERVENTIONS:
Behavioral: KITS Program — This is a 4-month psychosocial intervention for foster children entering kindergarten and their caregivers beginning the summer before kindergarten. The KITS intervention consists of: (a) child therapeutic play groups to facilitate the development of self-regulatory, social, and emergent literacy skills (2 times per week in summer, 1 times per week in the fall); (b) a bi-monthly psychoeducational support group to promote caregiver involvement in the child's emergent literacy and schooling and the use of effective parenting techniques; (c) home- and school-based behavioral consultation on an as needed basis.
  Other Names: Kids in Transition to School (KITS) Program
  Arms: KITS Program

SUMMARY:
The KITS project is a 5-year randomized trial to evaluate a program designed to enhance academic and social-emotional aspects of school readiness for foster preschoolers.

DETAILED DESCRIPTION:
The overarching goal of this research project is to conduct a randomized efficacy trial of a preventive intervention-the Kids in Transition to School (KITS) program-to enhance socioemotional and academic school readiness among preschool-aged foster children. Foster children are at great risk for poor social and academic school outcomes. Because of their experiences of early adversity, these children may have particular vulnerabilities that decrease the likelihood of a successful transition to school. Extensive prior research has shown that chronic early adversity is associated with alterations in the functioning of key neural systems (specifically, prefrontal cortex function and hypothalamic-pituitary-adrenal axis activity) related to self-regulation and stress reactivity. Alterations in these systems may interfere with children's abilities to relate to peers, to maintain focused attention, to follow directions, and to learn academic skills. Additionally, because these children are likely to have experienced multiple living transitions, they may be at a disadvantage in terms of caregiver involvement in school, a critical aspect of early school success. Foster children are recruited in the spring before they enter kindergarten and randomly assigned to the intervention and comparison conditions. The KITS intervention includes three components: (a) child therapeutic play groups to facilitate the development of self-regulatory, social, and emergent literacy skills; (b) a psychoeducational support group to promote caregiver involvement in the child's emergent literacy and schooling and the use of effective parenting techniques; (c) home- and school-based behavioral consultation. The intervention coincides with the transition into kindergarten. Multi-method, multi-agent assessments of the children's socioemotional readiness and literacy skills are conducted at baseline, kindergarten entry, and postkindergarten. We will examine the direct effects of the intervention on school readiness and kindergarten outcomes. We will also assess whether intervention effects are mediated through mechanisms of stress reactivity and regulation and caregiver variables. Finally, we will test for moderator effects of child and contextual characteristics including early adversity (prenatal/neonatal health, maltreatment history and placement history), child cognitive functioning, and placement transitions during the course of the study. An additional exploratory aim of the study is to examine intervention effects on first and second grade outcomes for subsamples of children. Group comparisons and longitudinal growth modeling will allow for evaluation of hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* a child currently in foster care
* living in Lane or Marion County, Oregon
* eligible to enter Kindergarten in fall of assessment year (age 5 by September 1 of assessment year)

Exclusion Criteria:

* medical or developmental condition which would prevent the child from completing the assessment tasks
* current or previous involvement in Oregon Social Learning Center treatment programs

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2005-09; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Early literacy skills | pre-intervention, pre-kindergarten, end of kindergarten
Social skills | pre-intervention, pre-kindergarten, end of kindergarten
Regulatory skills | pre-intervention, pre-kindergarten, end of kindergarten
Caregiver involvement | pre-intervention, pre-kindergarten, end of kindergarten

SECONDARY OUTCOMES:
Academic achievement | post-kindergarten, post 1st grade, post 2nd grade
Peer relations | post 1st grade, post 2nd grade

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Pears, PhD, Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Social Learning Center, Eugene, Oregon, United States

REFERENCES:
- [Background] Pears KC, Fisher PA, Bronz KD. An Intervention to Promote Social Emotional School Readiness in Foster Children: Preliminary Outcomes From a Pilot Study. School Psych Rev. 2007;36(4):665-673. PMID 19057655
- [Background] Pears KC, Fisher PA, Kim HK, Bruce J, Healey CV, Yoerger K. Immediate Effects of a School Readiness Intervention for Children in Foster Care. Early Educ Dev. 2013 Aug;24(6):771-791. doi: 10.1080/10409289.2013.736037. PMID 24015056
- [Background] Pears KC, Kim HK, Fisher PA. Effects of a School Readiness Intervention for Children in Foster Care on Oppositional and Aggressive Behaviors in Kindergarten. Child Youth Serv Rev. 2012 Dec;34(12):2361-2366. doi: 10.1016/j.childyouth.2012.08.015. No abstract available. PMID 23710106
- See also: Oregon Social Learning Center website — http://www.oslc.org